CLINICAL TRIAL: NCT01657695
Title: "Integrated Molecular/Imaging Technology for Characterization of Biological Aggressiveness of HCC in Patients Candidate to Liver Transplant"
Brief Title: Hepatocellular Carcinoma Growth and Molecular Aggressiveness
Acronym: UniRer
Status: Completed | Type: Observational
Sponsor: Prof. Facchinetti Fabio (Other)
Responsible Party: Sponsor-Investigator, Prof. Facchinetti Fabio, Clinical Professor, University of Modena and Reggio Emilia
Organization: University of Modena and Reggio Emilia (Other)
Other Study IDs: 10/08_CE_UniRer
Record Dates: First submitted 2012-07-29; First posted 2012-08-06 (Estimated); Last update posted 2012-10-02 (Estimated); Status verified 2012-09

CONDITIONS: Cirrhosis; Hepatocellular Carcinoma
Keywords: HCC; Computed tomography; Gene expression; Fractional growth
MeSH Terms: conditions — Fibrosis; Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We have designed custom arrays selecting those genes that, on the basis of literature and our own data, will be most informative regarding molecular pathways of relevance for HCC onset and progression and which have been already associated with decreased survival. These genes belong to cell cycle, apoptosis, cell proliferation, cell signaling, hypoxia and metastasis-prone pathways.
Oversight: Data Monitoring Committee: No

SUMMARY:
Our long-term objective is to develop a new tool based on a (molecular-biology) integrated imaging technology able to characterize and categorize hepatocellular carcinoma (HCC) patients in need of liver transplant (LT). To this end, our study aims at correlating specific imaging traits and fractional growth of individual tumors collected over a restricted time frame (T0 and at week 7 after first tumor detection), with a "molecular signature", obtained by custom microarray, histochemical and cytokine analysis. This should allow us to translate a series of purely morphologic information into a meaningful pathobiologic data sets. Validation of the integrated molecular-imaging tool will be performed prospectively by correlating the imaging-molecular data with HCC outcome in term of survival and disease-free survival after down staging procedures.

DETAILED DESCRIPTION:
Organ allocation in our region is regulated according to MELD score. Patients with hepatocellular carcinoma (HCC) receive an additional score depending on size of the tumor and the time spent in transplant waiting list. However, the advantage given to these patients is uniform and does not take into account the profound biological heterogeneity of individual HCCs. To make the additional score righteous, the investigators need to identify patients with aggressively growing HCC who require salvage transplantation while those with slow-growing HCC do not deserve the additional score.

All cirrhotics with suspect HCC identified at routine US screening will be therefore enrolled in the prospective imaging and bio-molecular study.

They will be subjected to two computed tomography (CT) exams at 7 weeks interval to define fractional tumor growth and imaging traits, baseline US-guided liver biopsy for microarray and histochemical characterization, serum sampling for cytokine assay. Survival, disease-free survival after downstaging and transplant outcome will be recorded and analyzed in relation with imaging and molecular data. The investigators expect to set up an accurate imaging and molecular diagnostic tool able to identify patients with aggressive HCC requiring urgent access to transplant, reliable in predicting survival, standardisable and not too expensive.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhotic patients at first US identification of a focal lesion compatible with HCC
* Age > than 18 years
* No contraindications to performance of CT
* No contraindications to performance of US-guided liver biopsy

Exclusion Criteria:

Patients will be excluded if

* are unable to give informed consent to the study;
* liver tissue obtained at biopsy is insufficient to perform molecular/histochemical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cirrhotic patients, at first diagnosis of HCC and potential liver transplant candidates
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2008-06; Primary Completion 2012-05 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Survival | 2 years
  Survival will be compared between patients with rapidly and slowly growing HCCs

SECONDARY OUTCOMES:
Response to therapy | 2 years
  Response to therapy (liver transplant, resection, TACE) will be compared between rapidly and slowly growing HCCs

CONTACTS AND LOCATIONS:
Overall Officials: Erica Villa, MD, Principal Investigator — University of Modena and Reggio Emilia
Locations (1):
- Azienda Ospedaliero-Universitaria, Modena, Italy

REFERENCES:
- [Derived] Critelli RM, Milosa F, Romanzi A, Lasagni S, Marcelli G, Di Marco L, Pivetti A, Schepis F, Romagnoli D, Mancarella S, Dituri F, Martinez-Chantar ML, Giannelli G, Villa E. Upregulation of the oestrogen target gene SIX1 is associated with higher growth speed and decreased survival in HCV-positive women with hepatocellular carcinoma. Oncol Lett. 2022 Sep 21;24(5):395. doi: 10.3892/ol.2022.13515. eCollection 2022 Nov. PMID 36276500
- [Derived] Villa E, Critelli R, Lei B, Marzocchi G, Camma C, Giannelli G, Pontisso P, Cabibbo G, Enea M, Colopi S, Caporali C, Pollicino T, Milosa F, Karampatou A, Todesca P, Bertolini E, Maccio L, Martinez-Chantar ML, Turola E, Del Buono M, De Maria N, Ballestri S, Schepis F, Loria P, Enrico Gerunda G, Losi L, Cillo U. Neoangiogenesis-related genes are hallmarks of fast-growing hepatocellular carcinomas and worst survival. Results from a prospective study. Gut. 2016 May;65(5):861-9. doi: 10.1136/gutjnl-2014-308483. Epub 2015 Feb 9. PMID 25666192